CLINICAL TRIAL: NCT03488017
Title: Evaluation of the Safety and Tolerability of an Ocular Coil
Brief Title: Ocular Coil Drug Delivery Comfort Trial
Acronym: OCDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 161042
Record Dates: First submitted 2018-03-19; First posted 2018-04-04 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Ocular Coil (left eye) (Experimental): Left eye
  Interventions: Device: Ocular Coil
- Placebo Ocular Coil (right eye) (Experimental): Right eye
  Interventions: Device: Ocular Coil

INTERVENTIONS:
Device: Ocular Coil — Non-invasive ocular device

SUMMARY:
The Ocular Coil is intended to provide drug delivery to the ocular surface. This study will evaluate the safety and tolerability of the placebo Ocular Coil in healthy subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and comfort of a placebo Ocular Coil for 28 days in 40 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Informed and having given informed consent
* Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

* Subjects with a history of eye disease that can make them vulnerable for irritation by the coil.
* Subjects wearing contact lenses (unless they are willing to replace them for glasses for the duration of the study).
* Subjects using eye drops (during the study).
* Subjects with an Oriental/Asian lid crease, because of their narrow fornix.
* Subjects who do not speak and/or write Dutch properly.
* Subjects with a history of serious adverse reaction or hypersensitivity to components of the ocular coil. or to ophthalmic anaesthetics
* Women who are pregnant or nursing their child, or have the intention to become pregnant during the course of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in terms of ocular irritation | 28 days
  Ocular irritation is assessed by slit lamp microscopy through evaluation of the ocular redness, inflammatory cells and flare.

SECONDARY OUTCOMES:
Total time of Ocular Coil retention | 28 days
  The total number of days that the Ocular Coil is worn by the participant (from placement until removal) is recorded.
Percentage of Participants in Each Response Category of Subject Comfort | 28 days
  Subject comfort is assessed via a custom-made questionnaire. This questionnaire includes several questions related to eye comfort (itchy feeling, foreign feeling, etc.) and uses a 5-point scale (from agree to do not agree) and a 4-point scale (from always to never). The percentage of participants in each response category is recorded.
Incidence of ocular adverse events | 28 days
  Incidence of ocular adverse events related to the Ocular Coil or the associated procedures (placement and removal) is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Hospital Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided